CLINICAL TRIAL: NCT00950300
Title: A Phase III, Randomized Open-Label Study to Compare the Pharmacokinetics, Efficacy, and Safety of Subcutaneous (SC) Trastuzumab With Intravenous (IV) Trastuzumab Administered in Women With HER2-Positive Early Breast Cancer (EBC)
Brief Title: A Study to Compare Subcutaneous (SC) Versus Intravenous (IV) Administration of Herceptin (Trastuzumab) in Women With Human Epidermal Growth Factor Receptor (HER) 2-Positive Early Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BO22227; 2008-007326-19 (EudraCT Number)
Record Dates: First submitted 2009-07-30; First posted 2009-07-31 (Estimated); Results first posted 2017-01-23 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2017-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Fluorouracil; Cyclophosphamide; Docetaxel; Epirubicin; Trastuzumab

ARMS (2):
- Herceptin IV + Chemotherapy (Active Comparator): Participants will receive Herceptin via IV infusion for 8 cycles prior to surgery and an additional 10 cycles after surgery. Docetaxel will be co-administered during Cycles 1 to 4; chemotherapy during Cycles 5 to 8 will include 5-fluorouracil, cyclophosphamide, and epirubicin. Herceptin IV will be given on Day 1 of each 21-day cycle, as 8 milligrams per kilogram (mg/kg) for a loading dose during Cycle 1 and as 6 mg/kg during subsequent cycles.
  Interventions: Drug: 5-Fluorouracil; Drug: Cyclophosphamide; Drug: Docetaxel; Drug: Epirubicin; Drug: Herceptin IV [trastuzumab]
- Herceptin SC + Chemotherapy (Experimental): Participants will receive Herceptin via SC injection for 8 cycles prior to surgery and an additional 10 cycles after surgery. Docetaxel will be co-administered during Cycles 1 to 4; chemotherapy during Cycles 5 to 8 will include 5-fluorouracil, cyclophosphamide, and epirubicin. Herceptin SC will be given on Day 1 of each 21-day cycle, as a 600-milligram (mg) fixed dose.
  Interventions: Drug: 5-Fluorouracil; Drug: Cyclophosphamide; Drug: Docetaxel; Drug: Epirubicin; Drug: Herceptin SC [trastuzumab]

INTERVENTIONS:
Drug: 5-Fluorouracil — Participants will receive 5-fluorouracil, 500 milligrams per meter-squared (mg/m^2) via IV bolus or infusion, on Day 1 of every 21-day cycle during Cycles 5 to 8.
Drug: Cyclophosphamide — Participants will receive cyclophosphamide, 500 mg/m^2 via IV bolus, on Day 1 of every 21-day cycle during Cycles 5 to 8.
Drug: Docetaxel — Participants will receive docetaxel, 75 mg/m^2 via IV infusion on Day 1 of every 21-day cycle during Cycles 1 to 4.
Drug: Epirubicin — Participants will receive epirubicin, 75 mg/m^2 via IV bolus or infusion, on Day 1 of every 21-day cycle during Cycles 5 to 8.
Drug: Herceptin IV [trastuzumab] — Herceptin will be administered as 8 mg/kg (loading dose during Cycle 1) and 6 mg/kg (subsequent cycles) via IV infusion on Day 1 of each 21-day cycle for a total of 18 cycles.
  Arms: Herceptin IV + Chemotherapy
Drug: Herceptin SC [trastuzumab] — Herceptin will be administered as fixed dose 600 mg SC on Day 1 of each 21-day cycle for a total of 18 cycles.
  Arms: Herceptin SC + Chemotherapy

SUMMARY:
In this open-label multicenter trial, participants with operable or locally advanced breast cancer will be randomized to pre-operative treatment with 8 cycles of chemotherapy (4 cycles of docetaxel followed by 4 cycles of 5-fluorouracil, epirubicin, and cyclophosphamide) concurrent with either SC Herceptin or IV Herceptin. After surgery, participants will receive a further 10 cycles of SC or IV Herceptin as per randomization to complete 1 year of treatment. All cycles will be 21 days in length. After the end of study treatment, participants will be followed for safety and efficacy for up to 5 years or until disease recurrence, whichever is earlier.

ELIGIBILITY:
Inclusion Criteria:

* Adult women greater than or equal to (≥) 18 years of age
* Non-metastatic primary invasive adenocarcinoma of the breast clinical stage I to IIIC, including inflammatory and multicentric/multifocal breast cancer, with tumor size ≥1 centimeter (cm) by ultrasound or ≥2 cm by palpation, centrally confirmed HER2-positive (immunohistochemical score [IHC] 3+ or in situ hybridization [ISH]-positive)
* At least 1 measurable lesion in breast or lymph nodes (≥1 cm by ultrasound or ≥2 cm by palpation), except for inflammatory carcinoma (T4d)
* Baseline left ventricular ejection fraction (LVEF) ≥55%
* Eastern Cooperative Oncology Group (ECOG) status of 0 or 1
* Adequate organ function at Baseline

Exclusion Criteria:

* History of any prior (ipsilateral and/or contralateral) invasive breast carcinoma
* Past or current history of malignant neoplasms, except for curatively treated basal and squamous cell carcinoma of the skin and in situ carcinoma of the cervix
* Metastatic disease
* Any prior therapy with anthracyclines
* Prior anti-HER2 therapy or biologic or immunotherapy
* Serious cardiac illness
* Pregnant or lactating women

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 596 (Actual)
Dates: Start 2009-10-16 (Actual); Primary Completion 2011-07-12 (Actual); Study Completion 2017-01-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (106):
- Argentina (2):
  - Centro Medico San Roque; Oncology Dept, San Miguel de Tucumán
  - Caipo; Oncology, San Miguel de Tucumán
- Brazil (8):
  - Hospital Sao Rafael - HSR, Salvador, Estado de Bahia
  - Hospital das Clinicas - UFPR; Quimioterapia, Curitiba, Paraná
  - Liga Norte Riograndense Contra O Câncer, Natal, Rio Grande do Norte
  - Clinica de Neoplasias Litoral, Itajaí, Santa Catarina
  - Hospital Amaral Carvalho, Jaú, São Paulo
  - Instituto do Cancer do Estado de Sao Paulo - ICESP, São Paulo, São Paulo
  - Hospital Perola Byington, São Paulo, São Paulo
  - Instituto de Oncologia de Sorocaba - CEPOS, Sorocaba, São Paulo
- Canada (2):
  - Hopital Maisonneuve- Rosemont; Oncology, Montreal, Quebec
  - CHU de Québec - Hôpital du Saint-Sacrement / ONCOLOGY, Québec
- Colombia (3):
  - Hospital Universitario San Ignacio, Bogotá
  - Grupo Salud Coop, Bogotá
  - Oncólogos de Occidente, Pereira
- Czechia (4):
  - Fakultni nemocnice Olomouc; Onkologicka klinika, Olomouc
  - Krajska Nemocnice Pardubice Neurologicka Klinika, Pardubice
  - Fakultni Thomayerova Nemocnice; Onkologicke Oddeleni, Prague
  - Lekarske Fakulty Univerzity Karlovy Fakultni Nemocnice Na Bulovce; Ustav Radiacni Onkologie, Prague
- Estonia (2):
  - North Estonia Medical Centre Foundation; Oncology Centre, Tallinn
  - Tartu University Hospital; Clinic of Hematology and Oncology, Tartu
- France (7):
  - HOPITAL JEAN MINJOZ; Oncologie, Besançon
  - Institut Daniel Hollard; Chimiotherapie Ambulatoire, Grenoble
  - Hopital Albert Michallon; Oncologie, La Tronche
  - Centre Jean Bernard, Le Mans
  - Hopital Saint Louis ; Service d Oncologie Medicale Fougere 6 (Pr Misset), Paris
  - Institut Jean Godinot; Hopital De Jour, Reims
  - Centre Rene Huguenin; Medecine B, Saint-Cloud
- Germany (10):
  - CAMPUS CHARITÉ MITTE; Tagesklinik für Onkologie u.Hämatologie, Berlin
  - Praxis Dr. Schoenegg, Berlin
  - Johanniter GmbH; Johanniter-Krankenhaus; Internistische Onkologie, Bonn
  - St. Johannes Hospital, Dortmund
  - Gynaekologisch-Onkologische Schwerpunktpraxis Prof. Dr. med. Lueck, Dr. Schrader und Dr. Noeding, Hanover
  - Sankt Elisabeth Krankenhaus; Gynaekology, Leipzig
  - Klinik Lippe Lemgo; Frauenklinik, Lemgo
  - Sana Klinikum Offenbach GmbH; Klinik für Gynäkologie & Geburtshilfe, Offenbach
  - Klinik Obergöltzsch; Abt. Gynäkologie, Rodewisch
  - Universitätsklinik Tübingen; Frauenklinik, Tübingen
- Centro Oncologico S.A., Guatemala City, Guatemala
- Queen Mary Hospital; Surgery, Hong Kong, Hong Kong
- Hungary (3):
  - Semmelweis Egyetem Onkologiai Központ, Budapest
  - Hospital of Aladar Petz; Dept of Oncoradiology, Győr
  - Szegedi Tudomanyegyetem, AOK, Szent-Gyorgyi Albert Klinikai Kozpont, Onkoterapias Klinika, Szeged
- Israel (2):
  - Hadassah Ein Karem Hospital; Oncology Dept, Jerusalem
  - Rabin Medical Center; Oncology Dept, Petah Tikva
- Italy (4):
  - Istituto Nazionale Tumori Irccs Fondazione g. Pascale;s.c. Ematologia Oncologica, Napoli, Campania
  - ASST DI CREMONA; Dip. Medicina - S.C. Oncologia, Cremona, Lombardy
  - Fondazione Salvatore Maugeri; Servizio Di Prevenzione Oncologica, Pavia, Lombardy
  - Fondazione Salvatore Maugeri, Pavia, Lombardy
- Mexico (2):
  - Hospital Privado San Jose; Oncologia, Obregón
  - Centro Oncológico Estatal; ISSSEMYM Oncología, Toluca
- Centro Oncologico America, Panama City, Panama
- Peru (5):
  - Hospital Nacional Carlos Alberto Seguin Escobedo-Essalud; Oncology & Haemathology, Arequipa
  - Hospital Nacional Edgardo Rebagliati Martins; Oncologia, Lima
  - Oncosalud Sac; Oncología, Lima
  - Unidad de Investigacion Oncologia Clinica - Piura; Unidad de Oncología Clínica, Piura
  - Clinica Ricardo Palma, San Isidro
- Poland (4):
  - Wojewodzki Szpital Zespolony; Oddział Onkologii, Elblag
  - COZL Oddzial Onkologii Klinicznej z pododdzialem Chemioterapii Dziennej, Lublin
  - Olsztyński Ośrodek Onkologiczny Kopernik sp. z o.o., Olsztyn
  - Centrum Onkologii - Instytut im. Marii Skłodowskiej-Curie Klinika Nowotworów Piersi i Chirurgii, Warsaw
- Russia (12):
  - FSBI"National Medical Research Center of Oncology named after N.N.Petrov" MHRF, Saint Petersburg, Sankt-Peterburg
  - Ivanovo Regional Oncology Dispensary, Ivanovo
  - Blokhin Cancer Research Center; Combined Treatment, Moscow
  - Moscow city oncology hospital #62 of Moscow Healthcare Department, Moscow
  - State Budget Institution of Healthcare of Stavropol region Pyatigorsk Oncology Dispensary, Pyatigorsk
  - SBI for HPE "Ryazan State Medical University n.a. I.P. Pavlov" of MoH of RF, Ryazan
  - Saint-Petersburg City Clinical Oncology Dispensary, Saint Petersburg
  - SBI of Healthcare Samara Regional Clinical Oncology Dispensary, Samara
  - Saratov Regional Clinical Hospital & Pathology Centre, Saratov
  - SBI of Healthcare of Stavropol region Stavropol Regional Clinical Oncology Dispensary, Stavropol
  - Tula Regional Oncology Dispensary, Tula
  - GUZ Vladimir Regional Clinical Oncological Dispensary, Vladimir
- Slovakia (2):
  - Vychodoslovensky onkologicky ustav, Košice
  - Nzz - Oncology Outpatient Clinic, Poprad
- South Africa (7):
  - National Hospital; Oncotherapy Dept, Bloemfontein
  - Cancercare, Cape Town
  - Groote Schuur Hospital ( Uni of Capetown ); Oncology Dept, Cape Town
  - Wits Donald Gordon Clinical Trial Centre; Medical Oncology, Parktown, Johannesburg
  - Pretoria-East Hospital; 1 Sanwood Park, Pretoria
  - Rondebosch Oncology Centre, Rondebosch
  - Sandton Oncology Centre, Sandton
- South Korea (4):
  - Gachon Medical School Gil Medical Center; Medical Oncology, Incheon
  - Samsung Medical Centre; Division of Hematology/Oncology, Seoul
  - Korea University Anam Hospital; Oncology Haemotology, Seoul
  - Asan Medical Center, Uni Ulsan Collegemedicine; Dept.Internal Medicine / Divisionhematology/Oncology, Seoul
- Spain (5):
  - Complejo Hospitalario Universitario de Santiago (CHUS) ; Servicio de Oncologia, Santiago de Compostela, LA Coruña
  - Hospital Universitari Sant Joan de Reus; Servicio de Oncologia, Reus, Tarragona
  - Hospital General Universitario Gregorio Marañon; Servicio de Oncologia, Madrid
  - Hospital Clinico Universitario de Valencia; Servicio de Onco-hematologia, Valencia
  - Hospital Universitario Miguel Servet; Servicio Oncologia, Zaragoza
- Sweden (2):
  - Skånes University Hospital, Skånes Department of Onclology, Lund
  - Akademiska sjukhuset, Onkologkliniken, Uppsala
- Taiwan (4):
  - Changhua Christian Hospital; Dept of Surgery, Changhua
  - Koo Foundation Sun Yat-Sen Cancer Center; Hemato-Oncology, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Medical Foundation-Taipei, Taoyuan District
- Thailand (5):
  - Chulalongkorn Hospital; Medical Oncology, Bangkok
  - National Cancer Inst., Bangkok
  - Phramongkutklao Hospital;Dept Surgery/Surgical Oncology Unit, Bangkok
  - Faculty of Med. Siriraj Hosp.; Med.-Div. of Med. Oncology, Bangkok
  - Prince of Songkla Uni ; Unit of Medical Oncology, Songkhla
- Turkey (Türkiye) (4):
  - Akdeniz University Medical Faculty; Medical Oncology Department, Antalya
  - Istanbul Uni of Medicine Faculty; Oncology Dept, Istanbul
  - Dokuz Eylul Uni Medical Faculty; Oncology Dept, Izmir
  - Hacettepe Uni Medical Faculty Hospital; Oncology Dept, Sıhhiye, Ankara

REFERENCES:
- [Derived] Jackisch C, Stroyakovskiy D, Pivot X, Ahn JS, Melichar B, Chen SC, Meyenberg C, Al-Sakaff N, Heinzmann D, Hegg R. Subcutaneous vs Intravenous Trastuzumab for Patients With ERBB2-Positive Early Breast Cancer: Final Analysis of the HannaH Phase 3 Randomized Clinical Trial. JAMA Oncol. 2019 May 1;5(5):e190339. doi: 10.1001/jamaoncol.2019.0339. Epub 2019 May 9. PMID 30998824
- [Derived] Ismael G, Hegg R, Muehlbauer S, Heinzmann D, Lum B, Kim SB, Pienkowski T, Lichinitser M, Semiglazov V, Melichar B, Jackisch C. Subcutaneous versus intravenous administration of (neo)adjuvant trastuzumab in patients with HER2-positive, clinical stage I-III breast cancer (HannaH study): a phase 3, open-label, multicentre, randomised trial. Lancet Oncol. 2012 Sep;13(9):869-78. doi: 10.1016/S1470-2045(12)70329-7. Epub 2012 Aug 9. PMID 22884505

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 833 participants were screened, out of which, 596 participants were enrolled into the study.
Groups:
- Herceptin IV + Chemotherapy: Participants received eight cycles of Herceptin IV plus chemotherapy prior to surgery and ten cycles of Herceptin IV after surgery. Chemotherapy consisted of docetaxel 75 milligrams per meter-squared (mg/m^2) every 21 days for four cycles followed by 5-fluorouracil 500 mg/m^2, epirubicin 75 mg/m^2, and cyclophosphamide 500 mg/m^2 (FEC) every 21 days for four cycles. Herceptin was administered as 8 milligrams per kilogram (mg/kg) on Day 1 and then as 6 mg/kg on Day 22 and every 21 days thereafter. The first eight cycles prior to surgery comprised the Neoadjuvant Treatment Period, and the ten cycles of Herceptin IV after surgery comprised the Adjuvant Treatment Period. Thereafter, participants entered the Treatment-Free Follow-Up (TFFU) Period. Participants who were withdrawn from the Neoadjuvant Treatment Period for any reason, or who experienced disease recurrence during either the Adjuvant Treatment Period or TFFU Period, could be entered into the Survival Follow-Up (SFU) Period.
- Herceptin SC + Chemotherapy: Participants received eight cycles of Herceptin SC plus chemotherapy prior to surgery and ten cycles of Herceptin SC after surgery. Chemotherapy consisted of docetaxel 75 mg/m^2 every 21 days for four cycles followed by FEC every 21 days for four cycles. Herceptin was administered as a 600-milligram (mg) fixed dose given every 21 days. The first eight cycles prior to surgery comprised the Neoadjuvant Treatment Period, and the ten cycles of Herceptin IV after surgery comprised the Adjuvant Treatment Period. Thereafter, participants entered the TFFU Period. Participants who were withdrawn from the Neoadjuvant Treatment Period for any reason, or who experienced disease recurrence during either the Adjuvant Treatment Period or TFFU Period, could be entered into the SFU Period.
Period: Neoadjuvant/Adjuvant Treatment Periods
Arm/Group | Herceptin IV + Chemotherapy | Herceptin SC + Chemotherapy
Started | 299 | 297
Received Neoadjuvant Treatment | 298 | 297
Underwent Surgery | 277 | 273
Entered Adjuvant Treatment | 277 | 274
Completed | 257 | 255
Not Completed | 42 | 42
Not completed — Adverse Event or Intercurrent Illness | 6 | 15
Not completed — Death | 1 | 3
Not completed — Insufficient Therapeutic Response | 3 | 0
Not completed — Violation of Selection Criteria | 2 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Participant Refusal/Withdrawal | 4 | 5
Not completed — Lost to Follow-up | 2 | 1
Not completed — Progression of Disease | 12 | 11
Not completed — Recurrence of Disease | 10 | 5
Not completed — Other | 1 | 1
Period: TFFU Period
Arm/Group | Herceptin IV + Chemotherapy | Herceptin SC + Chemotherapy
Started | 265 (Participants could withdraw from the study entirely or advance directly to the TFFU or SFU Period.) | 268 (Participants could withdraw from the study entirely or advance directly to the TFFU or SFU Period.)
Completed | 165 (Includes participants who completed either 2 years of follow-up or 5 years of follow-up.) | 161 (Includes participants who completed either 2 years of follow-up or 5 years of follow-up.)
Not Completed | 100 | 107
Not completed — Adverse Event or Intercurrent Illness | 3 | 4
Not completed — Death | 4 | 1
Not completed — Refused Treatment | 10 | 11
Not completed — Failure to Return | 16 | 16
Not completed — Recurrence of Disease | 63 | 72
Not completed — Other | 4 | 3
Period: SFU Period
Arm/Group | Herceptin IV + Chemotherapy | Herceptin SC + Chemotherapy
Started | 118 (Participants could withdraw from the study entirely or advance directly to the SFU Period.) | 123 (Participants could withdraw from the study entirely or advance directly to the SFU Period.)
Completed | 40 (Includes participants who completed either 2 years of follow-up or 5 years of follow-up.) | 45 (Includes participants who completed either 2 years of follow-up or 5 years of follow-up.)
Not Completed | 78 | 78
Not completed — Death | 44 | 42
Not completed — Lost to Follow-up | 30 | 28
Not completed — Withdrawal by Subject | 4 | 8

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Population: All participants with at least one efficacy assessment after administration of the first treatment cycle.
Groups:
- Herceptin IV + Chemotherapy: Participants received eight cycles of Herceptin IV plus chemotherapy prior to surgery and ten cycles of Herceptin IV after surgery. Chemotherapy consisted of docetaxel 75 mg/m^2 every 21 days for four cycles followed by FEC every 21 days for four cycles. Herceptin was administered as 8 mg/kg on Day 1 and then as 6 mg/kg on Day 22 and every 21 days thereafter. The first eight cycles prior to surgery comprised the Neoadjuvant Treatment Period, and the ten cycles of Herceptin IV after surgery comprised the Adjuvant Treatment Period. Thereafter, participants entered the TFFU Period. Participants who were withdrawn from the Neoadjuvant Treatment Period for any reason, or who experienced disease recurrence during either the Adjuvant Treatment Period or TFFU Period, could be entered into the SFU Period.
- Herceptin SC + Chemotherapy: Participants received eight cycles of Herceptin SC plus chemotherapy prior to surgery and ten cycles of Herceptin SC after surgery. Chemotherapy consisted of docetaxel 75 mg/m^2 every 21 days for four cycles followed by FEC every 21 days for four cycles. Herceptin was administered as a 600-mg fixed dose given every 21 days. The first eight cycles prior to surgery comprised the Neoadjuvant Treatment Period, and the ten cycles of Herceptin IV after surgery comprised the Adjuvant Treatment Period. Thereafter, participants entered the TFFU Period. Participants who were withdrawn from the Neoadjuvant Treatment Period for any reason, or who experienced disease recurrence during either the Adjuvant Treatment Period or TFFU Period, could be entered into the SFU Period.
- Total: Total of all reporting groups
Arm/Group | Herceptin IV + Chemotherapy | Herceptin SC + Chemotherapy | Total
Number analyzed (Participants) | 297 | 294 | 591
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.5 (10.83) | 50.3 (11.08) | 49.9 (10.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 297 | 294 | 591
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Observed Serum Trough Concentration (Ctrough) of Trastuzumab Prior to Surgery
Description: Pre-dose samples were obtained prior to surgery (Cycle 8). The observed Ctrough was recorded, averaged among all participants, and expressed in micrograms per milliliter (μg/mL).
Time Frame: Pre-dose (0 hours) on Day 1 of Cycle 8 (cycle length of 21 days)
Population: Primary Pharmacokinetic (PK) Per Protocol (PP) Population: All participants with at least one measurable trastuzumab serum concentration and who did not have any major protocol violations related to PK sampling for the primary endpoint.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Herceptin IV + Chemotherapy | Herceptin SC + Chemotherapy
Number analyzed (Participants) | 235 | 234
μg/mL | 57.8 (30.3) | 78.7 (43.9)
Statistical Analysis 1: Comparison: Herceptin IV + Chemotherapy vs Herceptin SC + Chemotherapy; PK sample size calculations based on percentage of coefficient of variation (CV%) for Ctrough of trastuzumab from previous metastatic breast cancer (MBC) and early breast cancer (EBC) studies. Because pre-surgery situation was comparable to MBC setting, interpatient CV% of 60 percent (%) was assumed and 130 participants per arm (260 participants total) were needed to demonstrate Ctrough comparability with 80% power if the true means of the two formulations did not differ by greater than (>) 5%; Test type: Non-Inferiority — Non-inferiority was concluded if the lower limit of the 90% confidence interval (CI) was greater than or equal to (≥) 0.8 for the geometric mean ratio; Geometric mean ratio = 1.33, 90% CI 2-sided [1.24 to 1.44] — Ratio of test treatment group (Herceptin SC + Chemotherapy) to reference treatment group (Herceptin IV + Chemotherapy)

2. Primary Outcome: Percentage of Participants With Pathological Complete Response (pCR)
Description: Participants were evaluated following eight cycles of treatment and after surgery to assess for pCR, defined as absence of neoplastic invasive cells in the breast according to pathologist examination. The percentage of participants with pCR was reported, and the 95% CI for one-sample binomial was constructed using the Pearson-Clopper method.
Time Frame: After surgery following eight cycles of Herceptin + chemotherapy (approximately 6 months from Baseline)
Population: Efficacy (E) PP Population: All participants with at least one on-treatment efficacy assessment who received a full eight cycles of study treatment according to randomization and who met additional protocol-specified criteria.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Herceptin IV + Chemotherapy | Herceptin SC + Chemotherapy
Number analyzed (Participants) | 263 | 260
percentage of participants | 40.7 [34.7 to 46.9] | 45.4 [39.2 to 51.7]
Statistical Analysis 1: Comparison: Herceptin IV + Chemotherapy vs Herceptin SC + Chemotherapy; Assuming pCR rates of at least 40% in both arms, 552 participants were necessary to conclude non-inferiority in pCR rate with a power of 80% using a one-sided 97.5% CI for the difference of the response rates and a non-inferiority margin of 12.5%; Test type: Non-Inferiority — Non-inferiority was concluded if the lower limit of the one-sided 97.5% CI was above -12.5% for the difference in response (pCR) rates; Difference in response rates = 4.70, 97.5% CI 1-sided [lower limit -4.0] — The one-sided 97.5% CI for the difference in response (pCR) rates was calculated using the Anderson-Hauck continuity correction

3. Secondary Outcome: Observed Ctrough of Trastuzumab After Surgery
Description: Pre-dose samples were obtained after surgery (Cycle 13). The observed Ctrough was recorded, averaged among all participants, and expressed in μg/mL.
Time Frame: Pre-dose (0 hours) on Day 1 of Cycle 13 (cycle length of 21 days)
Population: Secondary PKPP Population: All participants with at least one measurable trastuzumab serum concentration and who did not have any major protocol violations related to PK sampling for the secondary endpoint.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Herceptin IV + Chemotherapy | Herceptin SC + Chemotherapy
Number analyzed (Participants) | 223 | 227
μg/mL | 62.1 (37.1) | 90.4 (41.9)
Statistical Analysis 1: Comparison: Herceptin IV + Chemotherapy vs Herceptin SC + Chemotherapy; Additional supportive analysis; Test type: Other; Geometric mean ratio = 1.51, 90% CI 2-sided [1.40 to 1.63] — Ratio of test treatment group (Herceptin SC + Chemotherapy) to reference treatment group (Herceptin IV + Chemotherapy)

4. Secondary Outcome: Predicted Ctrough of Trastuzumab Prior to Surgery
Description: Predicted Ctrough at pre-dose prior to surgery (Cycle 8) was determined on the basis of a population PK model from Study BP22023 (NCT00800436). The mean predicted Ctrough was expressed in μg/mL.
Time Frame: Pre-dose (0 hours) on Day 1 of Cycle 8 (cycle length of 21 days)
Population: PKPP Population: All participants with at least one measurable trastuzumab serum concentration.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Herceptin IV + Chemotherapy | Herceptin SC + Chemotherapy
Number analyzed (Participants) | 276 | 278
μg/mL | 51.4 (19.4) | 80.3 (33.2)
Statistical Analysis 1: Comparison: Herceptin IV + Chemotherapy vs Herceptin SC + Chemotherapy; Additional supportive analysis; Test type: Other; Geometric mean ratio = 1.55, 90% CI 2-sided [1.46 to 1.64] — Ratio of test treatment group (Herceptin SC + Chemotherapy) to reference treatment group (Herceptin IV + Chemotherapy)

5. Secondary Outcome: Predicted Ctrough of Trastuzumab After Surgery
Description: Predicted Ctrough at pre-dose after surgery (Cycle 13) was determined on the basis of a population PK model from Study BP22023 (NCT00800436). The mean predicted Ctrough was expressed in μg/mL.
Time Frame: Pre-dose (0 hours) on Day 1 of Cycle 13 (cycle length of 21 days)
Population: PKPP Population; only participants with a Cycle 13 pre-dose PK measurement were included in the analysis.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Herceptin IV + Chemotherapy | Herceptin SC + Chemotherapy
Number analyzed (Participants) | 236 | 236
μg/mL | 51.7 (20.0) | 80.6 (33.4)
Statistical Analysis 1: Comparison: Herceptin IV + Chemotherapy vs Herceptin SC + Chemotherapy; Additional supportive analysis; Test type: Other; Geometric mean ratio = 1.55, 90% CI 2-sided [1.45 to 1.64] — Ratio of test treatment group (Herceptin SC + Chemotherapy) to reference treatment group (Herceptin IV + Chemotherapy)

6. Secondary Outcome: Number of Participants With Ctrough of Trastuzumab >20 μg/mL Prior to Surgery
Description: Pre-dose samples were obtained prior to surgery (Cycle 8). The number of participants who had an observed Ctrough >20 μg/mL was reported.
Time Frame: Pre-dose (0 hours) on Day 1 of Cycle 8 (cycle length of 21 days)
Population: Primary PKPP Population
Measure: Number; unit: participants
Arm/Group | Herceptin IV + Chemotherapy | Herceptin SC + Chemotherapy
Number analyzed (Participants) | 235 | 234
participants | 232 | 227

7. Secondary Outcome: Number of Participants With Ctrough of Trastuzumab >20 μg/mL After Surgery
Description: Pre-dose samples were obtained after surgery (Cycle 13). The number of participants who had an observed Ctrough >20 μg/mL was reported.
Time Frame: Pre-dose (0 hours) on Day 1 of Cycle 13 (cycle length of 21 days)
Population: Secondary PKPP Population
Measure: Number; unit: participants
Arm/Group | Herceptin IV + Chemotherapy | Herceptin SC + Chemotherapy
Number analyzed (Participants) | 223 | 227
participants | 216 | 227

8. Secondary Outcome: Maximum Serum Concentration (Cmax) of Trastuzumab Prior to Surgery
Description: PK samples were obtained prior to surgery (Cycle 7). The Cmax during Cycle 7 was recorded, averaged among all participants, and expressed in μg/mL.
Time Frame: Pre-dose (0 hours) and at end of 30-minute infusion (Herceptin IV only) on Day 1 of Cycle 7; on Days 2, 4, 8, 15 of Cycle 7; pre-dose (0 hours) on Day 1 of Cycle 8 (cycle length of 21 days)
Population: Primary PKPP Population; only those participants who provided evaluable data were included.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Herceptin IV + Chemotherapy | Herceptin SC + Chemotherapy
Number analyzed (Participants) | 235 | 233
μg/mL | 221 (118) | 149 (64.8)

9. Secondary Outcome: Time of Maximum Serum Concentration (Tmax) of Trastuzumab Prior to Surgery
Description: PK samples were obtained prior to surgery (Cycle 7). The Tmax during Cycle 7 was recorded, averaged among all participants, and expressed in days.
Time Frame: as for outcome 8
Population: Primary PKPP Population; only those participants who provided evaluable data were included.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Herceptin IV + Chemotherapy | Herceptin SC + Chemotherapy
Number analyzed (Participants) | 235 | 233
days | 0.05 (0.04) | 4.12 (2.91)

10. Secondary Outcome: Area Under the Concentration-Time Curve From 0 to 21 Days (AUC21d) of Trastuzumab Prior to Surgery
Description: PK samples were obtained prior to surgery (Cycle 7). Values were extrapolated beyond Day 15 to produce the area over the full 21-day cycle. The AUC21d value at Cycle 7 was calculated from trastuzumab concentration-time profiles using standard non-compartmental PK methods, averaged among all participants, and expressed in days multiplied by micrograms per milliliters (d*μg/mL).
Time Frame: as for outcome 8
Population: Primary PKPP Population; only those participants who provided evaluable data were included.
Measure: Mean (Standard Deviation); unit: d*μg/mL
Arm/Group | Herceptin IV + Chemotherapy | Herceptin SC + Chemotherapy
Number analyzed (Participants) | 235 | 233
d*μg/mL | 2056 (598) | 2268 (875)

11. Secondary Outcome: Cmax of Trastuzumab After Surgery
Description: PK samples were obtained after surgery (Cycle 12). The Cmax during Cycle 12 was recorded, averaged among all participants, and expressed in μg/mL.
Time Frame: Pre-dose (0 hours) and at end of 30-minute infusion (Herceptin IV only) on Day 1 of Cycle 12; on Days 2, 4, 8, 15 of Cycle 12; pre-dose (0 hours) on Day 1 of Cycle 13 (cycle length of 21 days)
Population: Secondary PKPP Population; only those participants who provided evaluable data were included.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Herceptin IV + Chemotherapy | Herceptin SC + Chemotherapy
Number analyzed (Participants) | 223 | 223
μg/mL | 230 (118) | 166 (58.8)

12. Secondary Outcome: Tmax of Trastuzumab After Surgery
Description: PK samples were obtained after surgery (Cycle 12). The Tmax during Cycle 12 was recorded, averaged among all participants, and expressed in days.
Time Frame: as for outcome 11
Population: Secondary PKPP Population; only those participants who provided evaluable data were included.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Herceptin IV + Chemotherapy | Herceptin SC + Chemotherapy
Number analyzed (Participants) | 223 | 222
days | 0.06 (0.13) | 4.08 (2.87)

13. Secondary Outcome: AUC21d of Trastuzumab After Surgery
Description: PK samples were obtained after surgery (Cycle 12). Values were extrapolated beyond Day 15 to produce the area over the full 21-day cycle. The AUC21d value at Cycle 12 was calculated from trastuzumab concentration-time profiles using standard non-compartmental PK methods, averaged among all participants, and expressed in d*μg/mL.
Time Frame: as for outcome 11
Population: Secondary PKPP Population; only those participants who provided evaluable data were included.
Measure: Mean (Standard Deviation); unit: d*μg/mL
Arm/Group | Herceptin IV + Chemotherapy | Herceptin SC + Chemotherapy
Number analyzed (Participants) | 223 | 223
d*μg/mL | 2179 (725) | 2610 (945)

14. Secondary Outcome: Percentage of Participants With Total Pathological Complete Response (tpCR)
Description: Participants were evaluated following eight cycles of treatment and after surgery to assess for tpCR, defined as absence of neoplastic invasive cells in the breast and axillary lymph nodes according to pathologist examination. The percentage of participants with tpCR was reported, and the 95% CI for one-sample binomial was constructed using the Pearson-Clopper method.
Time Frame: After surgery following eight cycles of Herceptin + chemotherapy (approximately 6 months from Baseline)
Population: EPP Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Herceptin IV + Chemotherapy | Herceptin SC + Chemotherapy
Number analyzed (Participants) | 263 | 260
percentage of participants | 34.2 [28.5 to 40.3] | 39.2 [33.3 to 45.5]
Statistical Analysis 1: Comparison: Herceptin IV + Chemotherapy vs Herceptin SC + Chemotherapy; Test type: Other; Difference in response rates = 5.01, 95% CI 2-sided [-3.5 to 13.5] — The 95% CI for the difference in response (tpCR) rates was calculated using the Anderson-Hauck continuity correction

15. Secondary Outcome: Percentage of Participants With Complete Response (CR) or Partial Response (PR) According to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.0, Among Those With Measurable Disease at Baseline
Description: Tumor response was assessed using RECIST version 1.0. CR was defined as disappearance of all target lesions and short-axis reduction of any pathological lymph nodes to less than (<) 10 millimeters (mm) with no prior assessment of progressive disease (PD). PR was defined as greater than or equal to (≥) 30% decrease from Baseline in sum diameter (SD) of target lesions with no prior assessment of PD. PD was defined as ≥20% relative increase and ≥5 mm of absolute increase in the SD of target lesions, taking as reference the smallest SD recorded since treatment started; or appearance of 1 or more new lesions. The percentage of participants with overall response of CR or PR at the end of neoadjuvant treatment was reported, and the 95% CI for one-sample binomial was constructed using the Pearson-Clopper method.
Time Frame: Tumor assessments at Baseline; on Day 1 of Cycles 3, 5, 7 (cycle length of 21 days); and at time of surgery following eight cycles of Herceptin + chemotherapy (approximately 6 months overall)
Population: EPP Population; only participants with measurable disease at Baseline were included.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Herceptin IV + Chemotherapy | Herceptin SC + Chemotherapy
Number analyzed (Participants) | 260 | 258
percentage of participants | 88.8 [84.4 to 92.4] | 87.2 [82.5 to 91.0]
Statistical Analysis 1: Comparison: Herceptin IV + Chemotherapy vs Herceptin SC + Chemotherapy; Test type: Other; Difference in response rates = -1.64, 95% CI 2-sided [-7.4 to 4.2] — The 95% CI for the difference in response (CR+PR) rates was calculated using the Anderson-Hauck continuity correction
Statistical Analysis 2: Comparison: Herceptin IV + Chemotherapy vs Herceptin SC + Chemotherapy; Test type: Other; Odds Ratio (OR) = 0.86, 95% CI 2-sided [0.50 to 1.46] — OR of test treatment group (Herceptin SC + Chemotherapy) to reference treatment group (Herceptin IV + Chemotherapy)

16. Secondary Outcome: Time to Response According to RECIST Version 1.0, Among Those With Measurable Disease at Baseline
Description: Tumor response was assessed using RECIST version 1.0. CR was defined as disappearance of all target lesions and short-axis reduction of any pathological lymph nodes to <10 mm with no prior assessment of PD. PR was defined as ≥30% decrease from Baseline in SD of target lesions with no prior assessment of PD. PD was defined as ≥20% relative increase and ≥5 mm of absolute increase in the SD of target lesions, taking as reference the smallest SD recorded since treatment started; or appearance of 1 or more new lesions. Time to response was defined as the time from first dose of study medication to the first assessment of CR or PR, which was the date the response was first documented by objective evidence, among participants with an overall response of CR or PR.
Time Frame: Tumor assessments at Baseline; on Day 1 Cycles 3, 5, 7 (cycle length of 21 days); and at time of surgery following eight cycles of chemotherapy (approximately 6 months overall)
Population: EPP Population; only participants with measurable disease at Baseline and a response of CR or PR were included.
Measure: Median (Full Range); unit: weeks
Arm/Group | Herceptin IV + Chemotherapy | Herceptin SC + Chemotherapy
Number analyzed (Participants) | 231 | 225
weeks | 6.14 [3 to 25] | 6.14 [3 to 28]

17. Secondary Outcome: Percentage of Participants Who Experienced a Protocol-Defined Event
Description: Protocol-defined events included disease recurrence/progression (local, regional, distant, contralateral) or death from any cause. Imaging was performed at specified visits for up to 5 years after last dose. Thereafter, participants were followed for survival only. The percentage of participants who experienced a protocol-defined event at any time during the study was reported.
Time Frame: Screening; Day 1 of Cycle 18 (cycle length of 21 days); and Months 6, 12, 24, 36, 48, 60 from last dose of Cycle 18; then every 6 months until withdrawal for any reason (up to approximately 87 months overall)
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Herceptin IV + Chemotherapy | Herceptin SC + Chemotherapy
Number analyzed (Participants) | 297 | 294
percentage of participants | 33.3 | 32.7

18. Secondary Outcome: Event-Free Survival (EFS)
Description: Protocol-defined events included disease recurrence or progression (local, regional, distant, contralateral) or death from any cause. Imaging was performed at specified visits for up to 5 years after last dose. Thereafter, participants were followed for survival only. EFS was estimated by Kaplan-Meier analysis and defined as the time from randomization to the first protocol-defined event.
Time Frame: as for outcome 17
Population: ITT Population
Measure: Median (Full Range); unit: months
Arm/Group | Herceptin IV + Chemotherapy | Herceptin SC + Chemotherapy
Number analyzed (Participants) | 297 | 294
months | NA [1 to 82] — The median time to event could not be determined because of a high number (>50%) of censored observations. Full range includes censored observations. | NA [1 to 76] — The median time to event could not be determined because of a high number (>50%) of censored observations. Full range includes censored observations.
Statistical Analysis 1: Comparison: Herceptin IV + Chemotherapy vs Herceptin SC + Chemotherapy; Test type: Other; p = 0.8651, Log Rank; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.74 to 1.29] — HR of test treatment group (Herceptin SC + Chemotherapy) to reference treatment group (Herceptin IV + Chemotherapy)

19. Secondary Outcome: Percentage of Participants Who Died
Description: The percentage of participants who died at any time during the study was reported.
Time Frame: Continuously during treatment (up to 12 months); at Months 1, 3, 6 from last dose of Cycle 18 (cycle length of 21 days); then every 6 months until withdrawal for any reason (up to approximately 87 months overall)
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Herceptin IV + Chemotherapy | Herceptin SC + Chemotherapy
Number analyzed (Participants) | 297 | 294
percentage of participants | 14.5 | 13.6

20. Secondary Outcome: Overall Survival (OS)
Description: OS was estimated by Kaplan-Meier analysis and defined as the time from randomization to death from any cause.
Time Frame: as for outcome 19
Population: ITT Population
Measure: Median (Full Range); unit: months
Arm/Group | Herceptin IV + Chemotherapy | Herceptin SC + Chemotherapy
Number analyzed (Participants) | 297 | 294
months | NA [2 to 82] — The median time to event could not be determined because of a high number (>50%) of censored observations. Full range includes censored observations. | NA [3 to 79] — The median time to event could not be determined because of a high number (>50%) of censored observations. Full range includes censored observations.
Statistical Analysis 1: Comparison: Herceptin IV + Chemotherapy vs Herceptin SC + Chemotherapy; Test type: Other; p = 0.7767, Log Rank; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.61 to 1.45] — HR of test treatment group (Herceptin SC + Chemotherapy) to reference treatment group (Herceptin IV + Chemotherapy)

21. Secondary Outcome: Number of Participants With Anti-Drug Antibodies (ADAs) Against Trastuzumab
Description: Participants provided PK samples for evaluation of anti-trastuzumab antibodies. The number of participants with "Treatment-induced ADAs" and "Treatment-enhanced ADA" against trastuzumab at any time during or after treatment was reported. Treatment-induced ADA = a participant with negative or missing Baseline ADA result(s) and at least one positive post-Baseline ADA result. Treatment-enhanced ADA = a participant with positive ADA result at Baseline who has one or more post Baseline titer results that are at least 0.60 titer unit greater than the Baseline titer result (four-fold increase of titer).
Time Frame: Baseline; pre-dose (0 hours) on Day 1 of Cycles 2, 5, 13, 18 (cycle length of 21 days); and Months 3, 6, 12, 18, 24, 30, 36, 42, 48, 54, 60 from last dose of Cycle 18
Population: Safety Population: All participants who received at least one dose of study medication. Here, Overall Number of Participants Analyzed = participants who were evaluable for this outcome measure.
Measure: Number; unit: participants
Arm/Group | Herceptin IV + Chemotherapy | Herceptin SC + Chemotherapy
Number analyzed (Participants) | 296 | 295
participants
  Treatment-induced ADAs | 28 | 46
  Treatment-enhanced ADA | 2 | 1

22. Secondary Outcome: Number of Participants With ADAs Against Recombinant Human Hyaluronidase (rHuPH20)
Description: Participants in the Herceptin SC arm provided PK samples for evaluation of anti-rHuPH20 antibodies. The number of participants with "Treatment-induced ADAs" and "Treatment-enhanced ADA" against rHuPH20 (an excipient unique to the SC formulation) at any time during or after treatment was reported. Treatment-induced ADA = a participant with negative or missing Baseline ADA result(s) and at least one positive post-Baseline ADA result. Treatment-enhanced ADA = a participant with positive ADA result at Baseline who has one or more post Baseline titer results that are at least 0.60 titer unit greater than the Baseline titer result (four-fold increase of titer).
Time Frame: as for outcome 21
Population: Safety Population; as rHuPH20 is unique to SC formulation, this outcome measure was applicable for "Herceptin SC + Chemotherapy" arm only. Here, Overall Number of Participants Analyzed = participants who were evaluable for this outcome measure.
Measure: Number; unit: participants
Arm/Group | Herceptin SC + Chemotherapy
Number analyzed (Participants) | 295
participants
  Treatment-induced ADA | 49
  Treatment-enhanced ADA | 13

ADVERSE EVENTS:
Time Frame: Approximately 87 months overall
Description: Analysis was performed on Safety Population.
Arm/Group | Herceptin IV + Chemotherapy | Herceptin SC + Chemotherapy
Serious Adverse Events (participants affected / at risk) | 45/298 | 65/297
Other Adverse Events (participants affected / at risk) | 277/298 | 283/297
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Herceptin IV + Chemotherapy (N=298) | Herceptin SC + Chemotherapy (N=297)
Respiratory tract infection viral (Infections and infestations) | 0 | 1
Lymphorrhoea (Vascular disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 2
Goitre (Endocrine disorders) | 1 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 10 | 13
Neutropenia (Blood and lymphatic system disorders) | 9 | 7
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 2
Pneumonia (Infections and infestations) | 4 | 2
Atypical pneumonia (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 2
Febrile infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
H1N1 influenza (Infections and infestations) | 1 | 0
Hepatitis B (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 2
Periorbital cellulitis (Infections and infestations) | 0 | 1
Postoperative wound infection (Infections and infestations) | 0 | 2
Respiratory tract infection (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 0 | 1
Abscess (Infections and infestations) | 0 | 1
Encephalitis viral (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Infected lymphocele (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Post procedural infection (Infections and infestations) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 2
General physical health deterioration (General disorders) | 0 | 1
Sudden death (General disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 1
Angina pectoris (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
Schizophrenia (Psychiatric disorders) | 0 | 1
Haematoma (Vascular disorders) | 1 | 1
Thrombophlebitis (Vascular disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 2 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Incision site haematoma (Injury, poisoning and procedural complications) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Pulmonary radiation injury (Injury, poisoning and procedural complications) | 0 | 1
Radiation pneumonitis (Injury, poisoning and procedural complications) | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dizziness (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 1
Ovarian haemorrhage (Reproductive system and breast disorders) | 0 | 1
Ovarian mass (Reproductive system and breast disorders) | 1 | 0
Vaginal prolapse (Reproductive system and breast disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour marker increased (Investigations) | 0 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 1
Mastitis (Infections and infestations) | 1 | 1
Tonsillitis bacterial (Infections and infestations) | 0 | 1
Death (General disorders) | 1 | 0
Ejection fraction (Investigations) | 0 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Breast abscess (Infections and infestations) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Herceptin IV + Chemotherapy (N=298) | Herceptin SC + Chemotherapy (N=297)
Alopecia (Skin and subcutaneous tissue disorders) | 188 | 187
Rash (Skin and subcutaneous tissue disorders) | 44 | 48
Nail disorder (Skin and subcutaneous tissue disorders) | 31 | 29
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 18 | 20
Pruritus (Skin and subcutaneous tissue disorders) | 27 | 26
Erythema (Skin and subcutaneous tissue disorders) | 8 | 21
Nausea (Gastrointestinal disorders) | 147 | 145
Diarrhoea (Gastrointestinal disorders) | 109 | 101
Vomiting (Gastrointestinal disorders) | 69 | 69
Stomatitis (Gastrointestinal disorders) | 51 | 57
Constipation (Gastrointestinal disorders) | 45 | 43
Dyspepsia (Gastrointestinal disorders) | 30 | 33
Abdominal pain upper (Gastrointestinal disorders) | 27 | 21
Abdominal pain (Gastrointestinal disorders) | 16 | 22
Asthenia (General disorders) | 75 | 75
Fatigue (General disorders) | 80 | 70
Mucosal inflammation (General disorders) | 39 | 31
Pyrexia (General disorders) | 35 | 35
Oedema peripheral (General disorders) | 30 | 23
Injection site pain (General disorders) | 0 | 18
Neutropenia (Blood and lymphatic system disorders) | 135 | 128
Leukopenia (Blood and lymphatic system disorders) | 46 | 30
Anaemia (Blood and lymphatic system disorders) | 41 | 34
Myalgia (Musculoskeletal and connective tissue disorders) | 54 | 61
Arthralgia (Musculoskeletal and connective tissue disorders) | 60 | 53
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 22 | 18
Back pain (Musculoskeletal and connective tissue disorders) | 25 | 26
Pain in extremity (Musculoskeletal and connective tissue disorders) | 26 | 29
Bone pain (Musculoskeletal and connective tissue disorders) | 10 | 19
Headache (Nervous system disorders) | 44 | 50
Peripheral sensory neuropathy (Nervous system disorders) | 27 | 33
Dysgeusia (Nervous system disorders) | 22 | 24
Dizziness (Nervous system disorders) | 28 | 29
Neuropathy peripheral (Nervous system disorders) | 18 | 24
Decreased appetite (Metabolism and nutrition disorders) | 59 | 58
Nasopharyngitis (Infections and infestations) | 40 | 24
Upper respiratory tract infection (Infections and infestations) | 30 | 30
Urinary tract infection (Infections and infestations) | 22 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 24 | 35
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 18 | 19
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 22 | 21
Incision site pain (Injury, poisoning and procedural complications) | 24 | 33
Procedural pain (Injury, poisoning and procedural complications) | 16 | 18
Radiation skin injury (Injury, poisoning and procedural complications) | 34 | 41
Hot flush (Vascular disorders) | 31 | 30
Hypertension (Vascular disorders) | 14 | 24
Insomnia (Psychiatric disorders) | 31 | 26
Alanine aminotransferase increased (Investigations) | 19 | 16
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 24 | 20
Dermatitis (Skin and subcutaneous tissue disorders) | 15 | 14
Oedema (General disorders) | 15 | 10
Pain (General disorders) | 15 | 12
Pharyngitis (Infections and infestations) | 11 | 15
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 19 | 19
Amenorrhoea (Reproductive system and breast disorders) | 10 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.